CLINICAL TRIAL: NCT06714487
Title: JUGUEMOS - Cognitive Stimulation Through Games : a New Active Aging Approach to Enhance Users' Everyday Challenges Sclerosis Multiple
Brief Title: Cognitive Stimulation in Patients With Sclerosis Multiple
Acronym: JuguEMos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IISPV-juguEMos-HTVC
Record Dates: First submitted 2015-11-23; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; play and Playthings; cognitive therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention): Neuropsychological evaluation including pre and 6 months without cognitive stimulation through games.
- Intervention with games (Experimental): Neuropsychological evaluation including pre and 6 months with cognitive stimulation three times a week through games.
  Interventions: Other: cognitive stimulation through games

INTERVENTIONS:
Other: cognitive stimulation through games — cognitive stimulation through games
  Arms: Intervention with games

SUMMARY:
The primary objective of the study is to determine if the training for 6 months with a specific set of games ( previously selected according to the cognitive domain stimulate : attention, memory , executive functions and processing speed ) , so improve significant neuropsychological performance of patients with Multiple Sclerosis Sender Recurrent ( RRMS ) and secondary progressive multiple sclerosis (SPMS ) , your mood and your quality of life.

Design : randomized clinical trial with a control group , coordinated a multicenter sample preselected patients.

DETAILED DESCRIPTION:
A total of 80 patients with RRMS or SPMS, which will be evaluated at baseline were included regarding various clinical, demographic, neuropsychological, psychometric and operational variables.

Subsequently patients will be randomized (in a ratio of 1: 1) to two groups different. The experimental group (EG = 40 patients) participate in a program of stimulation Cognitive group, while the control group (CG = 40 patients) did not receive any experimental intervention. All patients continue to receive drug treatment MS according to the standard treatment algorithms. At 6 months, once patients GE have completed treatment of cognitive stimulation, 80 patients will be reassessed respect to the same variables neuropsychological, psychometric and operation that had It has been evaluated at baseline.

Cognitive differences, clinics and operating both at baseline and at 6 be studied months among patients of GE responders and nonresponders to treatment stimulation cognitive and GC.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of RRMS or SPMS according to Poser criteria (1983) and McDonald (2001).
* Degree of disability between 1 ( clinical signs without disability) and 5.5 (capable of walk 100 meters without aid or rest , disability severe enough to prevent the activities of the whole ) day as the Disability Scale Kurtze (EDSS , 1983).
* Basic treatment for first-line MS ( immunomodulators).
* Complaints cognitive, functional gradation in the scale of dementia GDS ( Global Dementia Staging ) of Reisberg (1982 ) 2 and 4 .
* Patients who have mild to moderate cognitive impairment (have between 20 and 40 % of the altered neuropsychological tests).
* Signed informed consent .

Exclusion Criteria:

* Cognitive impairment associated with other medical diseases (Alzheimer's, stroke, Parkinson's disease, kidney disease, respiratory, hepatic, endocrine or hematological).
* Diagnosis of primary psychiatric disease with cognitive impairment in accordance with DSM-IV-TR criteria: schizophrenia, bipolar disorder, personality…
* Diagnosis or history of substance abuse or dependence.
* Score the Beck Depression Inventory II (BDI-II) greater than or equal to 30.
* Low Intelectual coeficient, inferred through obtaining a scale score less than 4 on the Vocabulary subtest of the WAIS-IV.
* Evidence of delusions, confusion or other disturbances of consciousness.
* Severe sensory deficits (visual and / or auditory)or functional illiteracy in which neuropsychological study can not be carried out.
* Patients treated with immunosuppressive drugs base or second line.
* Patients who are already receiving treatment or have cognitive rehabilitation received in the last 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Capacity to stimulate the functions cognitive, is why cognitive stimulation through strategies and neuropsychological specific set of board games, improve cognitive performance in patients with RRMS and PMSC . | Cognitive performance baseline (pre intervention) at 6 months (post intervention)
  Determine whether the training for 6 months with a specific set of table games (previously selected according to stimulate the cognitive domain: attention test score, memory test score, functions executive and processing speed test score, improved significantly, neuropsychological performance of patients with RRMS or SPMS questionnaires, their mood and quality of life, specify the measurement used with questionnaires. The project duration is 24 months.
  An intervention is applied for six months to two study groups. And it is expected to see a minimum difference of 1.5 points in the postintervention test scores.
  Phonetic verbal fluency test score; NEURONORMA project: words P in 1 minute). Subjects have to produce as many words as possible beginning with the letter P for 60 seconds. The total number of correct answers is analyzed, besides collecting errors and repetitions. WAIS-IV (score; is the number correctly coded from 0-133 in 120 seconds), HADS (score; from 0 to 21).

SECONDARY OUTCOMES:
Positive social interaction generated by the group reinforcement groups treatment will lead to improved mood of its participants. | Social interaction, baseline (pre intervention) at 6 months (post intervention)
  Positive social interaction generated by the group reinforcement groups treatment will lead to improved mood of its participants. The EVEA scale will measure mood states. (points of total score (10)).
Cognitive improvement achieved after participation in a group of cognitive stimulation through strategies and neuropsychological games, improve the quality of life Patients with RRMS and SPMS . | Quality of life (baseline, pre intervention) at 6 months (post intervention)
  Cognitive improvement as assessed by the MSQOL-54 scale (baseline, pre intervention) at 6 months (post intervention) at intervention group.
  The project duration is 24 months. Quality of life pre and post-intervention measured by Multiple Sclerosi Quality of Life MSQOL-54, is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. Quality of Life Questionnaire,: the total score obtained in the questionnaire will be recorded.
  Assessment of Quality of life through the following dimensions: physical functioning, role limitations due to physical problems, role limitations due to emotional problems, pain, emotional, fatigue or energy, perception of general health, social function and changes in health status. The total score obtained in the questionnaire will be recorded.